CLINICAL TRIAL: NCT01919333
Title: Anti-Mullerian Hormone Changes After Laparoscopic Ovarian Cystectomy for Endometrioma Compared With the Non-ovarian Conditions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Chamnan Tanprasertkul, Associate Professor, Thammasat University
Other Study IDs: MTU-OB-3-096/56
Record Dates: First submitted 2013-08-06; First posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Ovarian Reserve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- laparoscopic ovarian cystectomy: the group who laparoscopic ovarian cystectomy are performed for endometrioma
- laparoscopic non- ovarian pelvic surgery: the group whom laparoscopic non- ovarian pelvic surgery are performed

SUMMARY:
This aim of the study is to evaluate the impact of endometrioma and laparoscopic cystectomy on ovarian reserve as measured by serum antimullerian hormone and to study the different effects of levels of serum antimullerian hormone between laparoscopic cystectomy and the non-ovarian pelvic surgery.

ELIGIBILITY:
Inclusion Criteria:

* • Participants must be between the ages of 18 - 45 during enter the study .

  * Every participants have to completely understand the process of this study and have written informed consent .
  * Having regular menstrual cycles (21-35 days) at the time of operation
  * no evidence of any other endocrine disorders such as diabetes mellitus, thyroid dysfunction, hyperprolactinemia, congenital adrenal hyperplasia, Cushing's syndrome, or adrenal insufficiency.
  * undergo laparoscopic ovarian cystectomy or laparoscopic non- ovarian pelvic surgery for benign pelvic disease
  * No previous history of adnexal surgery
  * No any suspicious findings of malignant ovarian diseases
  * Never taking any medication such as oral pill and hormonal drugs within 3 months before the enrollment.
  * pathological diagnosis of excised ovarian tissue confirm as endometriotic cyst in study group and other benign pelvic disease in control group

Exclusion Criteria:

* polycystic ovarian syndrome according to the Rotterdam criteria

  * pathological report as the malignant diseases
  * have operation conversion to open-laparotomy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Reproductive women , age 18- 45 years who undergo laparoscopic ovarian cystectomy or laparoscopic non- ovarian pelvic surgery
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Serum AMH levels | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine , Thammasat university, Rangsit City Municipality, Pathumthanee, Thailand